CLINICAL TRIAL: NCT04289233
Title: Molecular & Cellular Characterisation of Oral Lichen Planus
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: RG_15-112
Record Dates: First submitted 2020-01-31; First posted 2020-02-28 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2021-04

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Unstimulated saliva Stimulated saliva Venous blood sample Surplus biopsy material
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The principal research objective is to provide enhanced understanding of the cellular and molecular events important in the pathogenesis of Oral Lichen Planus to enable improved diagnosis and development of novel treatments for patients.

DETAILED DESCRIPTION:
The following questions will also be addressed:

1. Are the histological architectural tissue changes that take place in oral lichen planus quantifiable using computer based imaging, graph theory and fractal geometry principles? Quantification of these changes would allow the development of a tool to facilitate the accurate measurement of response to treatment.
2. What is the nature of such architectural changes and what are the differences with normal, dysplastic and neoplastic epithelia (the investigators have morphometrical data collected from previous research to allow such comparisons).
3. Is it possible to produce evidence-based statistical classification into established diagnostic classes using the proposed methodology? This would contribute towards making histopathological diagnosis more quantitative, reproducible and accurate.
4. Is it possible to automate such morphometrical analysis/classification? This would allow large data sets to be screened automatically in a shorter time frame and at lower cost than human based screening.
5. Is it possible to determine differences in genetics and gene expression of keratinocytes involved in Oral Lichen Planus compared to those of 'normal' tissue by using biopsy material and an in vitro model of oral lichen planus?

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 16 years old or over
2. Patient is willing and able to provide valid informed consent
3. Patient is attending the Oral Lichen Planus clinic and will be having a routine clinical biopsy taken

Exclusion Criteria:

1. Patient under 16 years old
2. Patient is immunocompromised
3. Patients with comorbid disease state e.g. other inflammatory disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered at Birmingham Dental Hospital and attending a clinic for OLP diagnosis.
  Patients will be identified by their normal healthcare consultant and invited to participate.
  Informed consent will always be obtained prior to any study related procedures being undertaken.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-02-26 (Actual)

PRIMARY OUTCOMES:
Histological architecture | Through study completion, (maximum 12 months from the defined end of study)
  Are the histological architectural tissue changes that take place in oral lichen planus quantifiable using computer based imaging, graph theory and fractal geometry principles?
Comparisons with other dysplastic lesions | Through study completion, (maximum 12 months from the defined end of study)
  What is the nature of such architectural changes and what are the differences with normal, dysplastic and neoplastic epithelia
Statistical classifications | Through study completion, (maximum 12 months from the defined end of study)
  Is it possible to produce evidence-based statistical classification into established diagnostic classes using the proposed methodology
Automation of morphological features | Through study completion, (maximum 12 months from the defined end of study)
  Is it possible to automate such morphometrical analysis/classification?
Molecular expression of Oral Lichen Planus markers | Through study completion, (maximum 12 months from the defined end of study)
  Is it possible to determine differences in genetics and gene expression of keratinocytes involved in Oral Lichen Planus compared to those of 'normal' tissue by using biopsy material and an in vitro model of oral lichen planus?

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Landini, Phd, Principal Investigator — University of Birmingham
Locations (1):
- Birmingham Dental Hospital and School of Dentistry, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No